CLINICAL TRIAL: NCT02235155
Title: Mifepristone and Misoprostol for Mid-trimester Termination of Pregnancy (13-22 Weeks LMP) in Uzbekistan
Brief Title: Mifepristone and Misoprostol for Midtrimester Termination of Pregnancy in Uzbekistan
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Other Study IDs: 1017
Record Dates: First submitted 2014-08-29; First posted 2014-09-09 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Abortion in Second Trimester

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women of 13-22 weeks gestation: Pregnant women of 13-22 weeks gestation will receive 200 mg mifepristone followed 24-48 hours later by 400 mcg sublingual misoprostol every three hours until complete expulsion.

SUMMARY:
The primary goal is to examine the efficacy and feasibility of a mifepristone-misoprostol medical abortion regimen in terminating pregnancies 13-22 weeks in Uzbekistan.

ELIGIBILITY:
Inclusion Criteria:

* Meet legal criteria to obtain abortion
* Have an ongoing pregnancy of 13-22 weeks gestation
* Be willing to undergo a surgical completion if necessary
* Have no contraindications to study procedures, according to provider
* Be willing and able to consent to procedure, either by reading consent document or by having consent document read to her
* Be willing to follow study procedures

Exclusion Criteria:

* Known previous transmural uterine incision
* Known allergy to mifepristone or misoprostol/prostaglandin or other contraindications to the use of mifepristone or misoprostol
* Any contraindications to vaginal delivery, including placenta previa

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2014-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Proportion of abortions that are complete as a measure of efficacy | At 15 hours after the start of misoprostol administration
  It is a proportion that specifies how many abortions out of all initiated abortions are complete without recourse to surgical intervention within 15 hours after the start of misoprostol administration.

SECONDARY OUTCOMES:
Interval of time between induction with misoprostol to complete abortion | Every 3 hours from the start of misoprostol administration until complete abortion
  It is the length of time between the administration of the first dose of misoprostol and complete abortion.
Women's satisfaction with the method | At discharge, up to 5 days after enrollment
  It is a scale that assesses the level of a woman's satisfaction with the procedure.
Side effects experienced by women | Every 3 hours from the start of misoprostol administration until complete abortion
  It is a brief questionnaire that records all side effects experienced by women.
Pain experienced by women | At the time of discharge, up to 5 days after enrollment
  It is a scale that assesses the acceptability of pain experienced by the woman.
Complications during induction and after discharge | Every 3 hours from the start of misoprostol administration, up to 1 month after discharge
  It is a record of complications and their treatment during induction and up to 1 month after discharge.
Women's perception of acceptability of the procedure | At discharge, up to 5 days after enrollment
  It is a scale that assesses the acceptability of the procedure for the woman.
Provider's perception of acceptability of the method | At study completion, up to 2 years after study enrollment commences
  It is a questionnaire that assesses the acceptability of the method for the provider.
Total dose of misoprostol administered | Every 3 hours from start of misoprostol administration to complete abortion
  Count of the total dose of misoprostol administered from the first dose to complete abortion.

CONTACTS AND LOCATIONS:
Overall Officials: Dilfuza Kurbanbekova, PhD, MD, Principal Investigator — Women's Wellness Center, Uzbekistan; Tamar Tsereteli, PhD, MD, Principal Investigator — Gynuity Health Projects; Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (3):
- Uzbekistan (3):
  - Bukhara Maternity House No. 1, Bukhara
  - Samarkand Perinatal Center, Samarkand
  - Clinic No. 2, Tashkent Medical Academy, Tashkent

REFERENCES:
- [Derived] Platais I, Tsereteli T, Maystruk G, Kurbanbekova D, Winikoff B. A prospective study of mifepristone and unlimited dosing of sublingual misoprostol for termination of second-trimester pregnancy in Uzbekistan and Ukraine. BMJ Sex Reprod Health. 2019 Jun 4:bmjsrh-2018-200167. doi: 10.1136/bmjsrh-2018-200167. Online ahead of print. PMID 31164394